CLINICAL TRIAL: NCT03895281
Title: Clinical Evaluation of the FilmArray® Meningitis/Encephalitis (ME) Panel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Cao Qing, Director of Infectious Diseases, Shanghai Children's Medical Center
Other Study IDs: SCMC-ME
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Meningitis/Encephalitis
MeSH Terms: conditions — Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FilmArray Meningitis/Encephalitis (ME) Panel — The FilmArray ME pouch is a closed system disposable that houses all the chemistry required to isolate, amplify and detect nucleic acid from multiple meningitis and encephalitis pathogens within a single CSF specimen obtained from a lumbar puncture. The rigid plastic component (fitment) of the FilmArray ME pouch contains reagents in freeze-dried form. The flexible plastic portion of the pouch is divided into discrete segments (blisters) where the required chemical processes are carried out. The user of the FilmArray ME Panel loads the sample into the FilmArray ME pouch, places the pouch into the FilmArray instrument/Module, and starts the run. All other operations are automated.

SUMMARY:
The FilmArray Meningitis/Encephalitis (ME) Panel (hereinafter referred to as FilmArray ME Panel) is a qualitative multiplexed nucleic acid-based in vitro diagnostic test intended for use with FilmArray systems. The FilmArray ME Panel is capable of simultaneous detection and identification of multiple bacterial, viral, and yeast nucleic acids directly from cerebrospinal fluid (CSF) specimens obtained via lumbar puncture from individuals with signs and/or symptoms of meningitis and/or encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Residual cerebrospinal fluid samples after routine tests;
* Samples obtained by lumbar puncture;
* Sample volume is not less than 0.5 mL;
* Samples that have not been centrifuged;

Exclusion Criteria:

* Samples from repeatedly enrolled patients;
* Samples that have not been preserved as required

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with signs and/or symptoms of meningitis and/or encephalitis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of the FilmArray ME Panel | 6 days upon sample collection
  Percent Positive Agreement and Percent Negative Agreement between FilmArray Result and Comparator Assay

IPD SHARING:
Plan to Share IPD: Undecided